CLINICAL TRIAL: NCT03268278
Title: Efficacy of Buprenorphine on Postoperative Endodontic Analgesia
Acronym: EBPEA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of interest
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Thomas A. Montagnese, Associate Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHClevelandMCBupStudy
Record Dates: First submitted 2017-08-11; First posted 2017-08-31 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain
Keywords: analgesia; endodontic; postoperative
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Buprenorphine; Lidocaine; Epinephrine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- buprenorphine and local anesthetic (Active Comparator): buprenorphine added to local anesthetic
  Interventions: Drug: Buprenorphine; Drug: lidocaine, epinephrine (Local anesthetic)
- sterile saline and local anesthetic (Placebo Comparator): sterile saline (placebo) added to local anesthetic
  Interventions: Drug: Sterile saline; Drug: lidocaine, epinephrine (Local anesthetic)

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine plus local anesthetic
  Arms: buprenorphine and local anesthetic
Drug: Sterile saline — Placebo 1,8 ml
  Arms: sterile saline and local anesthetic
Drug: lidocaine, epinephrine (Local anesthetic) — 2% lidocaine 1:100,000 epinephrine

SUMMARY:
To see whether the addition of buprenorphone to local anesthesia will lengthen postoperative analgesia for endodontic pain

ELIGIBILITY:
Inclusion Criteria:

* persons with preoperative pain to percussion of a tooth with pulpal disease requiring endodontic therapy, healthy individuals, ASA Class I and II, no known allergies to the drugs being administered

Exclusion Criteria:

* pregnancy, allergy to buprenorphine, allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
The Efficacy of Buprenorphine in addition to Local Anesthetic in Providing Prolonged Postoperative Endodontic Analgesia | two years
  The number of patients with extended postoperative analgesia when compared to the baseline in pain scores on a visual analog scale during a three-day period will be analyzed. A questionnaire containing a visual analog scale and a log for recording the use of rescue analgesics will be used to gather the data.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No